CLINICAL TRIAL: NCT06970080
Title: Therapeutic Relevance of Abnormal Airway Morphology in Asthma: A Path to Optimized Management and Drug Development (AirPATH Study)
Brief Title: Therapeutic Relevance of Abnormal Airway Morphology in Asthma
Acronym: AirPATH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sarah Svenningsen, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Xe012
Record Dates: First submitted 2025-04-17; First posted 2025-05-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: asthma; computed tomography; corticosteroids; inhaled drug deposition; magnetic resonance imaging; airway morphology; eosinophilic inflammation
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Uncontrolled eosinophilic asthma (Experimental): In Phase I, participants will receive a doubling of their current ICS dose. If their asthma remains uncontrolled, they will receive an OCS burst in phase II.
  Interventions: Drug: Inhaled corticosteroid (ICS); Drug: Oral Corticosteroid (OCS)

INTERVENTIONS:
Drug: Inhaled corticosteroid (ICS) — In Phase I, participants will receive additional same dose of extra-fine particle ICS (i.e., their ICS would be doubled) for 12-weeks.
  Other Names: QVAR; hydrofloroalkaline-beclomethasone dipropionate
Drug: Oral Corticosteroid (OCS) — In phase II, participants will receive add-on oral prednisone (30mg/day) for one-week.
  Other Names: prednisone

SUMMARY:
Most individuals with asthma can effectively manage their symptoms and maintain normal lung function using inhaled medications, unfortunately, there is a subset of asthma sufferers whose symptoms, lung function, and risk of asthma attacks remain unimproved despite conventional inhaled medications. There could be several reasons for this. One possibility is that inhaled medications fail to reach the intended areas within the lungs, due to structural abnormalities within the airways themselves. Much like road conditions or closures can impede the speed and efficiency of vehicle travel, factors such as airway narrowing or mucus blockages, which are common in asthma, can obstruct the passage of inhaled medications through the airways. Our team has now optimized advanced medical imaging techniques, including magnetic resonance imaging (MRI) and computed tomography (CT), required to investigate this. This study will use these imaging methods to visually assess and measure individual patients' airways and determine whether abnormal airway structures impact how well they respond to inhaled and orally delivered medications. We anticipate finding that abnormal airway structures make inhaled medications less effective, but that they do not affect the response to oral medications.

DETAILED DESCRIPTION:
The cornerstone of asthma management lies in inhaled medications, including corticosteroids (ICS) and long-acting beta2-agonists (LABA). Unfortunately, individual responses to these first-line inhalers vary, and are ineffective in some people with asthma.

In asthma, the airways are the central site of disease pathology. Chronic airway inflammation, bronchial hyperresponsiveness, mucus plugging, and/or airway remodelling lead to luminal obstruction and airflow limitation that drive asthma symptoms. These factors can impact airflow, and the passage of inhaled drugs through the airways in asthma. Because optimal therapeutic effect likely depends, in part, on the dose topically deposited to the site of pathology, we propose that abnormal airway morphology may limit inhaled drug delivery to diseased airways and be a major factor contributing to poor response to inhaled drugs. Systemic (e.g., oral) drug delivery may achieve therapeutic targeting to diseased airways inaccessible by inhalation. This has not been investigated, and it constitutes the primary focus of the AirPATH study.

AirPATH is a two-phase open-label clinical study in adult patients with uncontrolled eosinophilic asthma to determine whether differences in their response to inhaled (ICS) and oral corticosteroid (OCS) treatments are predicted based on imaging-derived metrics of airway morphology and function.

Phase I Procedures Study Phase I is a 12-week clinical study of people with uncontrolled eosinophilic asthma. Patients will be screened for airway eosinophilia (sputum eosinophils ≥3% and/or FeNO ≥35ppb), uncontrolled asthma (ACQ-5 score ≥1.5), adequate inhaler technique and compliance. On clinical grounds, patients who meet these criteria require a "step-up" in their anti-inflammatory treatment. They will continue whatever ICS/LABA that they are on at screening and receive additional same dose of extra-fine particle ICS (i.e., their ICS would be doubled) for 12-weeks. Additional ICS will be delivered as equivalent of hydrofloroalkaline-beclomethasone dipropionate (Qvar) through a metered dose inhaler using an AeroChamber spacer. Patients will continue all their pre-study medication throughout the study.

Visit procedures: At screening (visit 1, week -1), demographics (age, biological sex, self-identified gender, BMI and race/ethnicity) and asthma characteristics will be collected (ICS dose, asthma duration), pre and post-bronchodilator pulmonary function tests (PFT) will be performed, sputum induction will be performed to quantify airway eosinophils, and the ACQ-5 will be completed to document asthma control. Eligible patients will proceed to a baseline visit (visit 2, week 0), and undergo inspiratory and expiratory chest CT, 129Xe and 1H MRI, PFTs, sputum induction, FeNO, blood draw, and complete questionnaires (ACQ-5, ACT, AQLQ), before their ICS dose is doubled. To determine the biological, physiological, and clinical response to additional ICS, patients will be followed-up at 12-weeks (visit 3) for outcome assessment, at which time all baseline (visit 2) procedures will be repeated.

Phase II Procedures Participants with persistent uncontrolled eosinophilic asthma (sputum eosinophils ≥3% and/or FeNO ≥35ppb and ACQ-5 score ≥1.5) after study Phase I will enter Phase II. Study phase II is a 1-week, clinical study in which all participants, regardless of their inhaled corticosteroid dose, will receive add-on oral prednisone (30mg/day) for one-week. Visit 3/week 12 will serve as the Phase II baseline, such that patients would have undergone inspiratory and expiratory chest CT, 129Xe and 1H MRI, PFTs, sputum induction, FeNO, blood draw, and completed the ACQ-5, before receiving add-on OCS. All other asthma medication would be continued. To document the biological, physiological, and clinical response to add-on OCS, participants will be followed-up at one-week (visit 4, week 13) for outcome assessment, at which time all baseline procedures except CT will be repeated.

Analysis Plan Multivariable linear regression models will be generated to determine if specific baseline imaging-metrics are independent predictors of biological response (∆ in sputum eosinophil percentage and FeNO), physiological response (∆ in 129Xe MRI VDP, FEV1, etc.), and/or clinical response (∆ in ACQ-5 score, etc.) to ICS (Phase I) and OCS (Phase II).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent.
* Able and willing to comply with the study protocol.
* Males and females ≥ 18 years of age.
* Asthma diagnosed by a respiratory physician.
* Airway hyperresponsiveness (defined as methacholine PC20 ≤8mg/mL) and/or bronchodilator reversibility (defined as post-bronchodilator FEV1 improvement ≥200mL and 12%) in the last 6 months
* ACQ ≥1.5 during the screening period.
* Sputum eosinophils ≥3% and/or FeNO ≥35ppb during the screening period.

Exclusion Criteria:

* Current smoker, defined as someone having smoked ≥1 cigarette/day (or vape/pipe/cigar/marijuana) for ≥30 days within 12 months prior to screening.
* Pregnant or breastfeeding
* Non-English speaking
* Oral corticosteroids in past 1-month
* Biologic therapy in past 6-months
* Unable to perform proper MDI technique during the screening period
* Other pulmonary diseases (e.g., chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis, pulmonary arterial hypertension, tuberculosis) requiring treatment within 12 months prior to screening.
* Unable to undergo MRI. Patient has an implanted mechanically, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist). Suffers from any physical, psychological, or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Biological response to additional ICS | 12 weeks
  Biological response to additional ICS evaluated as change from baseline in sputum eosinophil percent and FeNO at 12 weeks.
Biological response to add-on OCS | 1 week
  Biological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in sputum eosinophil percent and FeNO at one-week (Visit 4/Week 13).

SECONDARY OUTCOMES:
129Xe MRI ventilation defect percent (VDP) response to additional ICS | 12 weeks
  Change in 129Xe MRI VDP between baseline (week 0) and week 12.
FEV1 response to additional ICS | 12 weeks
  Physiological response to additional ICS evaluated as change from baseline in FEV1 at 12 weeks.
Respiratory system resistance (Rrs) at 5Hz response to additional ICS | 12 weeks
  Change in Rrs5Hz between baseline (week 0) and week 12.
Respiratory system reactance (Xrs) at 5Hz response to additional ICS | 12 weeks
  Physiological response to additional ICS evaluated as change from baseline in Xrs5Hz at 12 weeks.
Respiratory system resistance (Rrs) at 19Hz response to additional ICS | 12 weeks
  Physiological response to additional ICS evaluated as change from baseline in Rrs19Hz at 12 weeks.
Frequency dependence of Rrs (Rrs5-19Hz) response to additional ICS | 12 weeks
  Physiological response to additional ICS evaluated as change from baseline in Rrs5-19Hz at 12 weeks.
Integrated area of low frequency reactance (AX) response to additional ICS | 12 weeks
  Physiological response to additional ICS evaluated as change from baseline in AX at 12 weeks.
ACQ-5 response to additional ICS | 12 weeks
  Clinical response to additional ICS evaluated as change from baseline in Asthma Control Questionnaire-5 (ACQ-5) score at 12 weeks.
AQLQ response to additional ICS | 12 weeks
  Clinical response to additional ICS evaluated as change from baseline in Asthma Quality of Life Questionnaire (AQLQ) score at 12 weeks.
ACT response to additional ICS | 12 weeks
  Clinical response to additional ICS evaluated as change from baseline in Asthma Control Test (ACT) score at 12 weeks.
129Xe MRI ventilation defect percent (VDP) response to add-on OCS | 1 weeks
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in 129Xe MRI VDP at one-week (Visit 4/Week 13).
FEV1 response to add-on OCS | 1 week
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in FEV1 at one-week (Visit 4/Week 13).
Respiratory system resistance (Rrs) at 5Hz response to add-on OCS | 1 week
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in Rrs5Hz at one-week (Visit 4/Week 13).
Respiratory system reactance (Xrs) at 5Hz response to add-on OCS | 1 week
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in Xrs5Hz at one-week (Visit 4/Week 13).
Respiratory system resistance (Rrs) at 19Hz response to add-on OCS | 1 week
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in Rrs19Hz at one-week (Visit 4/Week 13).
Frequency dependence of Rrs (Rrs5-19Hz) response to add-on OCS | 1 week
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in Rrs5-19Hz at one-week (Visit 4/Week 13).
Integrated area of low frequency reactance (AX) response to add-on OCS | 1 week
  Physiological response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in AX at one-week (Visit 4/Week 13).
ACQ-5 response to add-on OCS | 1 week
  Clinical response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in the Asthma Control Questionnaire-5 (ACQ-5) score at one-week (Visit 4/Week 13).
AQLQ response to add-on OCS | 1 week
  Clinical response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in the Asthma Quality of Life Questionnaire (AQLQ) score at one-week (Visit 4/Week 13).
ACT response to add-on OCS | 1 week
  Clinical response to add-on OCS evaluated as change from Phase II baseline (Visit 3/Week 12) in the Asthma Control Test (ACT) score at one-week (Visit 4/Week 13).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: Undecided